CLINICAL TRIAL: NCT02867527
Title: Prospective Constitution of Database Gathering Data of Patients Suffering From Glaucoma Followed at University Hospital of Grenoble
Acronym: BDD_GLAUCOME
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC13.414
Record Dates: First submitted 2016-08-05; First posted 2016-08-16 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Few publications provide information on the natural history of glaucoma, outside of clinical trials do not always reflect what is observed in common situation for various reasons (specific selection criteria and sometimes restrictive, stronger motivations patients and physicians to comply with follow-up visits and prescribed treatments, etc.). Therefore, much information on the natural history of glaucoma are unknown to date (degradation rate of visual field and visual function over time, risk of blindness in the years following diagnosis, effects of various treatments to reduce intraocular pressure and preserving visual field deterioration, etc.). Obtaining such important data to improve the management of glaucoma patients (choice of treatment methods, identification of predictors of rapid change that can make choosing more aggressive treatment and more regular monitoring, etc.) requires the establishment of cohort of patients followed and treated with the methods usually used in current practice, and besides therapeutic trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is above 18 years
* Patients with primary or secondary glaucoma or both sides

Exclusion Criteria:

* Major person under guardianship or unable to consent
* Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data from all major subjects with primary or secondary glaucoma and examined for initial management or monitoring in the ophthalmology department of the University Hospital of Grenoble will be included in the database.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Degradation rate of visual field and visual function in patients treated with the methods usually used in current practice | 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No